CLINICAL TRIAL: NCT05477043
Title: Ultrasound Evaluation of Ureteral Patency After Uterosacral Ligaments Suspension
Brief Title: Ureteral Patency After Uterosacral Ligaments Suspension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: US-URETERS
Record Dates: First submitted 2022-05-03; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Uterovaginal Prolapse; Ureteral Injury; Surgery--Complications
Keywords: Uterovaginal prolapse; uterosacral ligament suspension; ureteral patency; ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group of study: Patients ≥ 18 years old subjected to uterosacral ligaments suspension surgical procedures for pelvic organs prolapse.
  Interventions: Diagnostic Test: Transabdominal ultrasound and cistoscopy

INTERVENTIONS:
Diagnostic Test: Transabdominal ultrasound and cistoscopy — Ultrasound detection of the bilateral ureteral jets vs absence of the ureteral jet on one side compared with the presence of bilateral ureteral jet on cystoscopy vs absence on one side.

SUMMARY:
Uterosacral ligament suspension (USLS) is a commonly performed procedure used to correct prolapse of the vaginal apex. The procedure consists of approximating the vaginal apex to the uterosacral ligaments with a series of sutures placed bilaterally, and is most often performed from a transvaginal approach. USLS is associated with favorable outcomes and is overall safe. However, given the anatomical proximity of the uterosacral ligaments to the ureters, ureteral injury during suspension suture placement may occur. Ureteral occlusion in this setting occurs as a result of partial or complete ligation, kinking or anatomical distortion by the nearby sutures. As a measure for avoiding these undesired sequelae, cystoscopy is usually performed after suspension suture placement during USLS to ensure visualization of bilateral ureteral flow. Any interruption of ureteral flow is usually addressed by removal of the suspension sutures, ureteral stenting, and, rarely, surgical repair of the ureter if severe injury is sustained.

Ultrasound can identify the ureteral jet of urine flowing into the bladder. Previous studies demonstrated ureteral jet asymmetry in case of obstruction, with an absent or weaker monolateral jet.

DETAILED DESCRIPTION:
It's a prospective observational monocentric study. 100 consecutive patients subjected to uterosacral ligaments suspension procedures for pelvic organs prolapse will be enrolled. Considering the surgical activity of our department we plan to enroll this number of patients within 18 months. After the surgical procedure, while still in the operatory room, they will be subjected to ultrasound evaluation of ureteral patency before being subjected to diagnostic cystoscopy. Ultrasound will be performed before cystoscopy in order not to be influenced by the results of the gold standard procedure. Ultrasound and cystoscopy will be performed by different operators in order not to be influenced by the results.

Intravenous somministration of 300 ml of saline solution will be performed 10 to 15 minutes before the end of the surgical procedure. Bladder will be filled with 300 ml of mannitol solution. All ultrasounds will be obtained with a convex 3.5-MHz probe. Ultrasound examination of the bladder will be performed in transverse planes. Bilateral simultaneous ureteral jet evaluation with power Doppler will be performed at the level of the ureterovesical junctions with a pulse repetition frequency set to detect low flow for 3 minutes, as previously described. The power Doppler field size will include the entire posterior wall of the bladder. Ureteral patency test will be considered normal if jets will be present at least once on each side. It will be considered abnormal when either absent or comparatively diminished on the ipsilateral side and well visualized on the contralateral side. It will be considered nondiagnostic when neither side was visualized during the 3 minutes. Ultrasound test results will be noted and after that diagnostic cystoscopy will be performed.

Postoperative care will be usual.

ELIGIBILITY:
Inclusion Criteria:

Patients ≥ 18 years old subjected to uterosacral ligaments suspension surgical procedures for pelvic organs prolapse.

Informed consent freely granted and acquired before the start of the study.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients subjected to uterosacral ligaments suspension procedures for pelvic organs prolapse will be enrolled.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Detection of ureteral patency | through study completion, an average of 1 year
  ultrasound detection of the bilateral ureteral jets vs absence of the ureteral jet on one side compared with the presence of bilateral ureteral jet on cystoscopy vs absence on one side.

SECONDARY OUTCOMES:
Duration | through study completion, an average of 1 year
  the duration of ultrasound procedure (minutes) compared with the duration of cystoscopy procedure (minutes).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Milano Bicocca, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: No